CLINICAL TRIAL: NCT00862680
Title: 4D PET/CT Imaging in Lung and Colorectal Cancer With Liver Metastasis
Brief Title: 4D PET/CT in Diagnosing Participants With Lung and Colorectal Cancer With Liver and Lung Metastasis
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2008-0853; NCI-2018-01858 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0853 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Malignant Neoplasm in the Liver; Metastatic Malignant Neoplasm in the Lung; Stage IV Colorectal Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic (4D PET/CT): Participants undergo 4D PET/CT scan over up to 12 minutes.
  Interventions: Procedure: 4-Dimensional Computed Tomography; Procedure: 4D PET Scan

INTERVENTIONS:
Procedure: 4-Dimensional Computed Tomography — Undergo 4D PET/CT
  Other Names: 4D Computed Tomography; 4DCT; Time-Resolved CT Data Acquisition
Procedure: 4D PET Scan — Undergo 4D PET/CT scan
  Other Names: 4D Gated PET; 4D Gated PET Scan; 4D PET

SUMMARY:
This trial studies how well 4 dimensional (D) positron emission tomography/computed tomography (PET/CT) works in diagnosing participants with lung or colorectal cancer that has spread to the liver and lung. Diagnostic procedures, such as PET/CT, may help find and diagnose disease and find out how far the disease has spread. But the motions made by breathing can reduce the image quality of the scan. Adjusting the scanner to 4D may allow for more breathing motion may improve the quality of the PET/CT images.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Study the impact of 4D positron emission tomography/computed tomography (PET/CT) imaging on the evaluation and staging of lung and colorectal cancer.

OUTLINE:

Participants undergo 4D PET/CT scan over up to 12 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected colorectal cancer with nodules in the lung or liver (1-2 cm in diameter) will be eligible for this study.
* Patients with suspected lung cancer with nodules in the lung or liver (1-2 cm in diameter) will be eligible for this study.

Exclusion Criteria:

* Patients that cannot tolerate being scanned for an additional 12 minutes with arms above their head will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-03-12 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-04-28 (Actual)

PRIMARY OUTCOMES:
Maximum lesion standardized uptake value (SUVmax) for gated and ungated positron emission tomography/computed tomography (PET/CT) scans | Up to 10 years
  Will be compared using a one-sided paired t-test.
Impact of the difference in SUVmax on the lesion detectability and staging of the evaluated patients | Up to 10 years
  two nuclear medicine physicians will assess the impact of the difference in SUVmax on the lesion detectablility and staging of the evaluated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Mawlawi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org